CLINICAL TRIAL: NCT05312684
Title: The Relationship Between Anticholinergic Burden and Postoperative Complications After Cardiac Surgery in Older Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bilal Katipoglu, M.D, Gulhane Training and Research Hospital
Other Study IDs: 22-2476
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High anticholinergic burden: ACB scale score 1 or >1 as a high anticholinergic buden
  Interventions: Procedure: cardiac surgery
- Normal anticholinergic burden: ACB scale score <1 as a control group
  Interventions: Procedure: cardiac surgery

INTERVENTIONS:
Procedure: cardiac surgery — cardiovascular surgery including valve repair/replacement or CABG or combined procedures

SUMMARY:
Drugs with anticholinergic properties are widely prescribed in the elderly population, despite increasing evidence in the literature regarding side effects and adverse outcomes. As is known, many drugs have anticholinergic activity, which means that they block the binding of the neurotransmitter acetylcholine to the muscarinic receptor. In this case, the occurrence of anticholinergic side effects becomes inevitable. Central effects such as cognitive impairment, dizziness, sedation, confusion or delirium, and peripheral effects such as dry mouth, dry eyes, constipation, urinary retention, and tachycardia begin to be seen in patients. Anticholinergic load refers to the cumulative effect of taking one or more drugs with anticholinergic activity. This cumulative effect is a strong indicator of cognitive and physical deterioration, especially in the elderly population. It is also associated with adverse outcomes such as falls, impaired functioning, and higher rates of hospitalization and death.

Anticholinergic load scales include scales that facilitate the work of physicians used in clinical practice to predict anticholinergic side effects in humans. Although there are many different scales used at this point, one of the scales with the highest validity and reliability in recent studies are Anticholinergic cognitive burden scale (ACB) and Anticholinergic risk scale (ARS). To the best of our knowledge, we could not find any study on postoperative complications, length of hospital stay and mortality after cardiac surgery with these scales. Therefore, we aimed to examine the relationship between possible complications after cardiac surgery and anticholinergic load scales showing the cumulative effect of preoperative drugs.

ELIGIBILITY:
Inclusion Criteria:

* It is planned to include patients over the age of 65 who underwent cardiac surgery in the research population.
* Gender discrimination will not be considered.

Exclusion Criteria:

* Those who are under the age of 65,
* Those who have non-cardiac surgery,
* Those whose drug records cannot be accessed

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: It is planned to include patients over the age of 65 who underwent cardiac surgery in the study population.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complication | 1 month fellow-up
  Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Katipoglu, Principal Investigator — Gulhane Training and Research Hospital
Locations (1):
- Gulhane training and research hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Katipoglu B, Kurtbeyoglu S, Demir ZA, Mavioglu HL. The effect of the anticholinergic burden on mortality following elective cardiac surgery. Curr Med Res Opin. 2024 Jan;40(1):27-34. doi: 10.1080/03007995.2023.2288278. Epub 2024 Jan 3. PMID 37999982